CLINICAL TRIAL: NCT04494854
Title: Perceptions, Representations and Experiences of Malaria Prophylaxis in Patients Born in Endemic Areas and Living in France.
Acronym: PREPAP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: PREPAP
Record Dates: First submitted 2020-07-17; First posted 2020-07-31 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Malaria; Disease, Infectious; Travel-Associated Infections
Keywords: perception, representation, experience, questionnaire
MeSH Terms: conditions — Malaria; Communicable Diseases; Travel-Related Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to analyze the perceptions, representations and expe-riences of malaria prophylaxis in patients born in endemic areas and living in France.

This analysis could lead to better understanding and communication between the medical profession and patients in malaria. It would also provide patient-specific responses to their expectations, as to their families.

DETAILED DESCRIPTION:
Malaria is the most common vector-borne (mosquito-borne) disease in the world. It is caused by a parasite called Plasmodium, and is transmitted to humans by an Anopheles mosquito bite. Malaria rages in most intertropical regions and in 91 countries. Hence, almost half of the world's population is expose. The estimated number of cases was 219 million (CI95 = 203-262) in 2018, including 200 million in Africa (92%). The number of deaths in 2017 reached 435,000, of which 93% in Africa.

In 2018, in metropolitan France, the National Reference Center recorded 2,730 reported cases including one case of indigenous malaria, the other cases were import cases. There were 12.8% of severe forms and 84.9% of the patients were of African origin and had stayed in Africa, without taking anti-malaria chemoprophylaxis.

The fight against malaria is therefore a major public health issue in the world and in France, with in particular the need for better access to pre-trip consultations, in town or in hospital, and improved key messages deliverance on this frequent and potentially serious pathology, and also the means of protection (chemoprophylaxis, repellents and mosquito nets). The role of general practitioners is essential in this fight since they represent the first source of information for 60% of patients.

To this effect, Recommendations for good practice for the management of imported malaria actualized and published in 2018 emphasizes these preventive measures for travelers bound for endemic areas.

The non-compliance rate was estimated at 29% in a 2007 study by Pistone et al. in patients from endemic areas when they are among the most affected patients. These data have not yet been verified for more than 10 years, and it seems important to actualized this knowledge in the light of social changes.

In addition, prevention methods borrowed from herbal medicine are sometimes offered elsewhere, such as Artemisia herbal teas, despite the scientific data that caused a lack of effectiveness.

Overall, few studies have explored the reasons for this obstacle to chemoprophylaxis and classically proposed anti-vector measures and a better understanding could allow a better delivery of information during our consultations.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Born in malaria endemic areas and living in France
* Having malaria or not
* Ready for no opposition for participation in the protocol

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients unable to give free and informed consent
* Patients under judicial protection

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be offered to patients born in endemic areas and living in France.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Identify perceptions, representations and experiences of malaria prophylaxis in patients coming from endemic areas living in France. | Through study completion, an average of 30 minutes
  The semi directive interview

SECONDARY OUTCOMES:
Identification of dialogue tools allowing a better relationship of trust between doctor and patient within the framework of a prevention consultation, and better delivery of key information | Through study completion, an average of 30 minutes
  The main themes identified through thematic coding will be used to develop the basis for a medical speech expected by patients and adapted to their needs

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier intercommunal de Villeneuve St Georges, Villeneuve-Saint-Georges, France